CLINICAL TRIAL: NCT06584916
Title: A Phase 3b, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Orforglipron Once Daily Versus Placebo for Maintenance of Body Weight Reduction in Participants Who Have Obesity or Overweight With Weight-Related Comorbidities
Brief Title: A Study of Orforglipron for the Maintenance of Body Weight Reduction in Participants Who Have Obesity or Overweight With Weight-Related Comorbidities (ATTAIN-MAINTAIN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27239; J2A-MC-GZPN (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Overweight
Keywords: Maintenance; Weight maintenance; Body weight changes; Weight loss; Incretins; Hormones; Hormone substitutes; Hormone antagonists; Physiological effects of drugs
MeSH Terms: conditions — Obesity; Overweight; Body Weight Changes; Weight Loss | interventions — orforglipron

STUDY DESIGN:
Intervention Model Description: Phase 3b
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orforglipron (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Placebo (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Arms: Orforglipron
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of orforglipron on maintenance of body weight reduction.

DETAILED DESCRIPTION:
All enrolled participants will have completed SURMOUNT-5 (I8F-MC-GPHJ; NCT05822830) on treatment and meet further eligibility and randomization criteria. All endpoints for this study will be evaluated separately per each intervention arm of SURMOUNT-5.

ELIGIBILITY:
Inclusion Criteria:

* Have completed the SURMOUNT-5 study on study treatment

Exclusion Criteria:

* Have Type 1 Diabetes, Type 2 Diabetes, or any other types of diabetes, history of ketoacidosis, or hyperosmolar state/coma
* Have a prior or planned surgical treatment for obesity
* Have acute or chronic hepatitis
* Have a history of acute or chronic pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Percent Maintenance of Body Weight Reduction Achieved in SURMOUNT-5 | Week 52

SECONDARY OUTCOMES:
Percent Change from SURMOUNT-5 Baseline in Body Weight Prior to Start of Treatment | Week 52
Number of Participants Maintaining ≥80% of the Body Weight Reduction Achieved in SURMOUNT-5 | Week 52
Change from Baseline in Body Weight | Baseline, Week 52
Change from Baseline in Waist Circumference | Baseline, Week 52
Percent Maintenance of Body Weight Reduction Achieved in SURMOUNT-5 | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (29):
- United States (27):
  - Cahaba Research, Birmingham, Alabama
  - Cahaba Research - Pelham, Pelham, Alabama
  - Southern California Dermatology, Inc., Santa Ana, California
  - Encompass Clinical Research, Spring Valley, California
  - University Clinical Investigators, Inc., Tustin, California
  - New Horizon Research Center, Miami, Florida
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - L-MARC Research Center, Louisville, Kentucky
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Prime Health and Wellness/SKYCRNG, Fayette, Mississippi
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - Palm Research Center Sunset, Las Vegas, Nevada
  - Weill Cornell Medical College, New York, New York
  - PharmQuest Life Sciences, LLC, Greensboro, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - WR-Clinsearch, LLC, Chattanooga, Tennessee
  - The University of Texas Health Science Center at Houston, Bellaire, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
- Puerto Rico (2):
  - Puerto Rico Medical Research, Ponce
  - Wellness clinical Research Vega Baja, Vega Baja

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/